CLINICAL TRIAL: NCT05181436
Title: A Cross- Sectional Study on the Prevalence of Malaysian Children Aged ≥ 6 to ≤ 36 Months at Risk of Anaemia
Brief Title: The Prevalence of Malaysian Children Aged ≥ 6 to ≤ 36 Months at Risk of Anaemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Danone Specialized Nutrition (M) Sdn Bhd (Industry)
Responsible Party: Sponsor
Other Study IDs: MD21-002
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Anemia
Keywords: anaemia; paediatrics
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Malaysian children aged ≥ 6 months to ≤ 36 months: The study population consists of Malaysian children aged ≥ 6 months to ≤ 36 months seen at Mother and Child Health Clinic (MCHC).
  Interventions: Diagnostic Test: measuring Total Haemoglobin (SpHb) using Masimo Rad-67.

INTERVENTIONS:
Diagnostic Test: measuring Total Haemoglobin (SpHb) using Masimo Rad-67. — To determine the prevalence of Malaysian children aged ≥ 6 to ≤ 36 months at risk of anaemia by measuring Total Haemoglobin (SpHb) using Masimo Rad-67.

SUMMARY:
The main purpose of this study is to determine the prevalence of Malaysian children aged ≥ 6 to ≤ 36 months at risk of anaemia by measuring Total Haemoglobin (SpHb) using a non-invasive haemoglobin assessment. Eligible subjects, and their parent(s) / legally acceptable representative(s) where applicable, who fulfil all the inclusion and none of the exclusion criteria will be enrolled into the study. Parameters will be recorded during the subjects visit at the MCHC using a self-administered 24-hour Diet Recall. Demographics and subject / family characteristics will be recorded at this visit by using questionnaire built into Iron Strong app which act as a data collection tool.For subjects with haemoglobin level <12 g/dL, the subject will be considered "at risk of anaemia" and as a standard operating procedure, the child will be referred to HCPs for further clinical assessment.

DETAILED DESCRIPTION:
Eligible subjects, and their parent(s) / legally acceptable representative(s) where applicable, who fulfil all the inclusion and none of the exclusion criteria will be enrolled into the study. Recruitment at the study sites will continue until required number subjects have been enrolled.

Parameters will be recorded during the subjects visit at the MCHC. Parent(s) / legally acceptable representative(s) will be asked to report subject dietary intake using a self-administered 24-hour Diet Recall. A Site Research Assistant will be present to assist with the completion of the 24-hour Diet Recall.

Demographics and subject / family characteristics will be recorded at this visit by using questionnaire built into Iron Strong app. The Iron Strong app, as a data collection tool includes an optical character recognition (OCR) model that allows user (by taking a picture) to accurately predicts all units and digits on Masimo Rad-67 device and store the data within the app / server. The access of the application is only possible via email invitation to Site Investigator / Research Assistant.

Masimo Rad-67 is a non-invasive device for total haemoglobin screening. A clip with sensor attached to Masimo Rad-67 will be place on the child's finger / toe, reading will take approximately 30 seconds.

For subjects with haemoglobin level <12 g/dL, the subject will be considered "at risk of anaemia" and as a standard operating procedure, the child will be referred to HCPs for further clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient children aged ≥ 6 months to ≤ 36 months at MCHC accompanied by their primary caretaker who could be parents/ grandparents / relatives.
2. Written consent from parent(s) / grandparents / relatives / legally acceptable representative(s) who are the primary caretaker of the child, who themselves are aged ≥18 years, to consent and comply with the terms and conditions of the study.

Exclusion Criteria:

1. Children with any medical condition that, in the opinion of the Investigator, would not be suitable for enrolment into the study. The examples of such medical condition include: severe chromosome / genetic abnormalities, severe neurological disorders which may cause feeding difficulties, severe congenital heart disease, severe acute malnutrition, gastrointestinal disorders that result in malabsorption (e.g. coeliac disease), malignancies, and any other medical condition in which the Investigator considers that interventions to increase nutritional intake may not be effective in improving weight gain and nutritional status.
2. Children participating in any other studies involving iron fortified foods / supplementation.
3. Parent(s) / legally acceptable representative(s) who have insufficient ability to understand or communicate in English and / or Bahasa Malaysia and / or Chinese (Mandarin).

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of Malaysian children aged ≥ 6 months to ≤ 36 months seen at Mother and Child Health Clinic (MCHC). A sample size of 1200 will be required after accounting for 10% each of screen failures and dropouts. Any withdrawn subjects /screen failures will be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Malaysian Children aged ≥ 6 to ≤ 36 months with SpHb (g/dL) <12 g/dL vs ≥12 g/dL measured using Masimo Rad-67. | 6 months
  Percentage of Malaysian Children aged ≥ 6 to ≤ 36 months with SpHb (g/dL) <12 g/dL vs ≥12 g/dL measured using Masimo Rad-67.

SECONDARY OUTCOMES:
Mean Haemoglobin among Malaysian children aged ≥ 6 to ≤ 36 months. Proportion of Malaysia children aged ≥ 6 to ≤ 36 months with SpHb (g/dL) < 11g/dL vs ≥11g/dL measured using Masimo Rad-67. | 6 months
  Mean Haemoglobin among Malaysian children aged ≥ 6 to ≤ 36 months. Proportion of Malaysia children aged ≥ 6 to ≤ 36 months with SpHb (g/dL) < 11g/dL vs ≥11g/dL measured using Masimo Rad-67.
Socio-demographic characteristics of child and parent(s) assisted and administered by Site Investigator. | 6 months
  Socio-demographic characteristics of child and parent(s) assisted and administered by Site Investigator.
Dietary intake using self-administered 24-hour Diet Recall interviewed and recorded by RA / Site Investigator. | 6 months
  Dietary intake using self-administered 24-hour Diet Recall interviewed and recorded by RA / Site Investigator.
Height / Length & weight recorded by RA / Site Investigator for their corresponding WHO Weight for Age, Height for Age Z-Scores for data analysis. | 6 months
  Height / Length & weight recorded by RA / Site Investigator for their corresponding WHO Weight for Age, Height for Age Z-Scores for data analysis.
Correlation between nutritional status (WHO Z-Scores, Total Energy intake / day, Protein intake / day, Iron intake / day) and risk of anaemia among Malaysian children aged ≥ 6 to ≤ 36 months. | 6 months
  Correlation between nutritional status (WHO Z-Scores, Total Energy intake / day, Protein intake / day, Iron intake / day) and risk of anaemia among Malaysian children aged ≥ 6 to ≤ 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Yazid Jalaludin, Principal Investigator — Department of Paediatrics, University Malaya Medical Centre
Locations (1):
- Department of Paediatrics, University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
This study is an industry sponsored research. Danone Specialized Nutrition (Malaysia) Sdn Bhd being the sponsor of the research is the exclusive owner of the study data as mutually agreed in the Clinical Trial Agreement. Investigators can be part of publication team and author of the manuscript as mutually agreed in the Clinical Trial Agreement.
  Proposals from Investigators for access to additional study data research,manuscript writing, knowledge sharing, reporting to ministries etc purposes can be given with permission by Danone Malaysia when applicable.